CLINICAL TRIAL: NCT04607369
Title: Implementation of the NEDS EyeCTester App and NEDS Server Analysis Software Into the Homes of Patients With Neuro-ophthalmic, Retinal and Other Diseases to Enhance Early Detection of Active Eye Disease.
Brief Title: Implementation of the NEDS EyeCTester App
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Neuro-Eye Diagnostic Systems, LLC (Industry)
Collaborators: Neuro-ophthalmology of Texas PLLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20190049
Record Dates: First submitted 2020-10-07; First posted 2020-10-29 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Optic Nerve Disease; Macular Disease; Visual Pathway Disorder
Keywords: Amsler Grid; Visual Field Defects; 10-2 Visual Field; Optic Nerve Diseases; Macula Diseases; Visual Pathway Disorders; Vision Monitoring
MeSH Terms: conditions — Optic Nerve Diseases; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (7):
- Groups in General all were done under the wcgIRB, even those that were Practice groups: Groups 1-3 were practice groups, gathering smartphone app installation, functional and usability feedback in preparation for later phase groups
  Groups 4a and 4b Cohort 1 and 2 is the FDA application finalized and submitted study groups
  Group 5-6 currently in continuing clinical trial during FDA application process
  Interventions: Device: EyeCTester
- 1-3,5 Developmental team(1), Technician(2) and Non-Clinical Groups(3) 5. Retinal practice: Individuals on the developmental team, staff members and outside clinic people 5 Retinal Practice (to do after FDA approval)
  Interventions: Device: EyeCTester
- 4a. Cohort 1. FDA group: Patients in Neuro-Ophthalmology of Texas (NOT) PLLC practice which has referrals from multiple practices including retinal patients.
  Interventions: Device: EyeCTester
- 4b. Cohort 2. FDA group: Patients in NOT practice
  Interventions: Device: EyeCTester
- 6 At Home use of app in continuing clinical trial during FDA decision: Patients are educated on the app at home via app video clips and brochure, and as necessary, online training with COA (ophthalmic assistants/technicians or other trained educators) in order to do remote physiologic vision monitoring or preclinic near vision check.
  Interventions: Device: EyeCTester
- 7a Cohort 1 FDA group responding to AI: Normal patients were tested with standard near vision tests compared with the smartphone app near vision tests. All patients were trained at home with app videos and by COA via telemedicine before coming to clinic.
  Interventions: Device: EyeCTester
- 7b Cohort 2 FDA group responding to AI: Normal patients were tested with standard near vision tests compared with the smartphone app near vision tests. All patients were trained at home with app videos and by COA via telemedicine before coming to clinic.
  Interventions: Device: EyeCTester

INTERVENTIONS:
Device: EyeCTester — Smartphone app that allows vision testing

SUMMARY:
Group 4a and 4b was an FDA trial that showed that patients who have an Amsler grid abnormality on paper, have a similar abnormality on the app.

Group 7a and 7b was an FDA trial that showed that normal patients do not have false positives on the Amsler app as well as on the Amsler paper version. Further Vision on the app is slightly better than vision on the standard Sloan near card using a formula (vision is 7/10th of a line better on the app).

DETAILED DESCRIPTION:
Detailed Description of 4A and 4B: A series of patients with central visual defects were identified and their names were given to the unblinded clinical coordinator. The clinical coordinator contacted the patients, described the study, arranged the appointments to come to the clinic one-at-a-time for a dedicated visit to participate in the study. Each patient experienced the same study process for their visit:

1. Met with the unblinded Clinical Coordinator who had the patient sign the informed consent after detailed explanation.
2. Had the Clinical Coordinator put a number tag on the patient, and this was the number that the blinded participants of the study were to use for these subjects. Additionally, random numbers were used on the test forms.
3. Patients met with blinded test trainer where the patient was provided standardized instruction for use of Amsler grid on-paper test, the Amsler grid on EyeQTester device, visual acuity and color sensitivity on paper and on the device. The instruction was enhanced between Cohort 1 and Cohort 2 as approved by the IRB for the different instruction protocol (see below discussion). Also, patients were given a test which they must pass in order to enter the trial.
4. Patients then met with the blinded test administrator where the patient took the tests with no coaching. The test admin confirmed that the environmental parameters were similar across all patients over the course of the study.
5. The patient completed test and re-test sequences.
6. All test results with assigned random numbers were reported by the test administrator to the Clinical Coordinator who provided batches of blinded results to the Data Coordinator.

The investigators knew from prior clinic experience that the patients required a new and more detailed educational experience than was standard in order to have more reliable results for both the paper and app Amsler Grid test, in order to measure the central visual fields. The investigators focused on carefully training the patient through both written material and a video where the educational administrator was there to review this with the patient. The education focused on:

1. What are "defects" and how to identify and report them.
2. How to draw the above defects with attention to distance from the fixation point, size of the defect as well as its density.

Training enhancement was prompted midway through the trial, when the unblinded sponsor and clinical coordinator reviewed patient test results. Initial conclusion was that the patients exhibited defect identification on both paper and app that could possibly be enhanced by improving the educational protocol. An updated educational protocol was provided which the sponsor discussed with the educational team which was implemented to test if this updated patient education would result in more reliable results. It was decided to utilize updated educational approach for all patients on both paper and the app. Additionally, the investigators, added a stylus for the app (replacing the patient's finger) in order to more closely simulate a pen which is utilized for the paper. This updated approach was submitted and approved by the IRB.

As a result of the above, a decision was made to have two cohorts in the study, the early education cohort 1 and the later education cohort 2. Patients in cohort 1 were trained on the device to draw a defect on the screen with the tip of their finger but on paper to use a pen. Patients in cohort 2 were trained on the device to draw a defect on the screen with a stylus and on paper with a pen. The result in Cohort 2 was that consistency of the patients test results were better for both test and re-test for both the Amsler grid on-paper and the EyeCTester device.

The statistical analysis in this report shows the overall results and also the improved results in Cohort 2 that likely is attributed to these educational enhancement and stylus additions.

The full protocol for the trial including the training is available in the WIRB trial documentation.

Sample Size Calculation by our statistician was verified to be the sample size used was statistically acceptable.

Summary: Amsler app and paper version were equivalent, and best when using a stylus on the app.

Detailed Description of 7A and 7 B A series of patients 22 and over without any vision problems being examined similar to the above (see WIRB description) with a different education protocol consisting of in-home video on the app, telemedical connection by COA to confirm teaching was understood, and if not reteach.

The statistical analysis in this report shows the overall results showed that the vision testing standard and app were similar, with better vision tested on the app, by a formula that approximates, 7/10 of a line better.

The statistical analysis in this report shows the overall results showed that the color testing standard and app were similar.

The statistical analysis in this report shows the overall results showed that the Amsler grid testing via standard near vision tests and app were exactly the same with neither having false positives.

The full protocol for the trial including the training is available in the WIRB trial documentation.

Sample Size Calculation by our statistician was verified to be the sample size used was statistically acceptable.

ELIGIBILITY:
Inclusion Criteria for 4a and 4b:

The participant must have at least one eye which complies with all the inclusion criteria

Inclusion criteria:

1. Patients have had a standard ICNVT in the last six months which could potentially qualify a patient's eye for study participation. This information will be used to determine whether to proceed with screening the patient with the remaining study selection criteria below.
2. In the proposed study eye, the patient has at least one scotoma or field-cut, metamorphopsia or doubling area that is non-overlapping and that has boundaries separated by more than 1 degree (the appendix describes "degree" measurements more fully). This means that if there are many scotoma's or areas of metamorphopsia or doubling, all but one is overlapping, the one that is not overlapping with required separation does qualify for the trial, while the others do not.
3. Age 18 or above 18 years old was selected as the minimum age because this study is only intended to evaluate patients who will follow directions well and can sign the consent alone.
4. If the patient uses corrective lenses, then if needed we will provide patients with an ophthalmologist configured optical trial lens frame with lenses configured to provide their near vision correction at 16 inches. We do this to eliminate the effect of multifocal or progressive lens viewing issues at near (from viewing through the wrong portion of the lens) on testing results. In a future study, potentially in this same trial, we may examine the effect of personal lenses on testing results. The patient must be able to tolerate wearing the optical trial frame without discomfort or problems viewing in these lenses.
5. Able to perform a short test provided in the clinic to measure if the patient can work with both the paper Amsler Grid as well as the Smart-phone Amsler grid. This test will be evaluated with standardized review and scoring by the Educator of the patient's performance, which will require an 80 percent score or better. The idea of this test is to be certain the combination of cognitive, motor and visual abilities of the patient is at the level that can easily for hold the paper grid (on a small clipboard) as well as hold the smart-phone in hand and for both modalities be steady enough to understand how to draw and to be able to draw on the paper and smart-phone Amsler grid per directions of the Educator. The provided iPhone 6 is technically similar to recent smart-phone models and demonstrates ease of use as tested by our team.
6. Visual acuity is to be no worse than 20/80 (LogMAR +0.50) at a viewing distance of 16 inches. At this distance the letter size will be 1.86 mm tall.
7. The patient must have the ability to directly focus on a 2.5 mm fixation point. This target is the size of the 20/80 Sloan optotype (LogMAR +0.50). In this fashion we can mostly ensure that direct, rather than eccentric viewing is performed. Eccentric viewing is not optimum for this trial as it may interfere with test repeatability if the eccentric viewing patient is not consistently using the same portion of their eye to view the test. Were this the case, the scotoma/field-cut positions may vary. It is acceptable for a scotoma or a field-cut to impinge on the fixation point as long as the density of the scotoma or a field-cut does not prevent direct viewing of the fixation point. The Eye Examiner EE (including the ophthalmologist and educator) will monitor and document whether the patient appears to be using direct visualization of the chart.
8. The patient's eyes should not be dilated.
9. The patient should have a static ophthalmic condition as determined by the sponsor that is not causing pain or discomfort and is not expected to change in the short timeframe between tests. Patients with recent eye surgery, should be stable as documented by Q & A with patient's eye care provider or in the patient's medical record if access is available.

Exclusion Criteria:

The participant must have at least one eye which complies with none of the exclusion criteria listed below.

1. A normal Amsler Grid with no scotoma or field-cut. Patients without Amsler defects are not the intended population of this study.
2. Before the education session, should the patient exhibit cognitive, motor problem (weakness, tremor, ataxia, etc.) or visual problems that prevent the patient from independently performing one or more of the near vision tests via the standard ICNVT or via SPNVT as described above in item 5 of Inclusion criteria.
3. Dilation of either eye on the day of and day prior to the trial examination because it limits accommodation as well as may increase in light sensitivity.
4. In the study eye, a scotoma or field-cut that is larger than 90% of the Amsler grid (90 cm2 or 360 squares).
5. In the study eye, the patient has scotomas or field-cuts, all of which are smaller than 0.0013% of the Amsler grid (0.13 cm2 or 1/2 of one Amsler grid square). Such small sized scotomas or field-cuts may reduce drawing accuracy on both Amsler Grid tests and may be undetectable on the 10-2.
6. Overlapping scotomas or field-cuts to all the scotomas present, because they add complexity to the study without adding value to the study results.
7. Two or more unreliable Visual Field test results. During the study, patient's visual field, will be tested using the Zeiss Humphrey® Field Analyzer 10-2 which will produce a "Single Field" outcome that includes reliability indices. The HFA 10-2 measurement to be carried out using the SITA standard test and the standard Goldmann III stimulus size. Only reliable VFs to be used in the analyses, defined as a fixation loss (FL) rate < 20% and a false-positive (FP) rate < 15%, following the manufacturer's recommendation for SITA measurements.
8. Should the patient appear to have unreliable parameters by 10-2 testing with one test, this test will not be evaluated, however, should the second 10-2 test be reliable, this test will be used to compare with the Amsler Grid results.

Study Criteria for Group 7

Age Limits:22 and over

1. Inclusion Criteria for 7A and 7B:

   * Must be 22 years old or older.
   * Have already been seen or will be seen by an optometrist or ophthalmologist.
   * Have normal vision as defined as best corrected vision of 20/20 or better.
   * Have a normal posterior pole OCT.
   * Have signed the informed consent.
2. Exclusion Criteria:

   * Patients younger than 22
   * Have a visual acuity worse than 20/20
   * Have macula pathology based on an abnormal posterior pole OCT exam
   * Have conditions that can interfere with Amsler grid testing for example tremors, trouble focusing, due to moving eyes (nystagmus) or trouble with concentration (e.g., ADDH) or cognition problems, based on known diagnoses in the chart or if history is obtained of these conditions during enrollment.
   * Individuals who fail the test in the office after training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For FDA approval Cohort 4a and 4b are the 2 groups being evaluated.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-01-09 (Estimated); Study Completion 2023-01-09 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure for Groups 4a and 4b: | Study was conducted for each patient in one day.
  The Test-Retest Repeatability for the identified three common near-vision procedures will be measured to determine sample sizes to reach the objectives of this study.
  Patients will be recruited from a neuro-ophthalmology and/or retina clinic's new or established patient population. Thirty willing patients with known Amsler grid abnormalities (metamorphopsia, scotoma, field-cut field-cut) will each complete the study protocol. Test results will be statistically analyzed to compare the app test with the in-office paper test versions. This analysis will allow the population size to be measured which is needed for valid test results.
Secondary Outcome Measure for Groups 4a and 4b | Study was conducted for each patient in one day.
  The limits of agreement will be reported by comparing the difference in measurements taken using In Clinic Near Vision Tests (ICNVT) vs Smart Phone Near Vision Tests (SPNVT). The investigators will determine the 95% limits of agreement by calculating the mean difference between ICNVT and SPNVT as well as the standard deviation. Histograms will be used to verify that the data is normally distributed. If the data is not normally distributed appropriate statistical transformation will be made by working directly with ratios.
  Once population size is determined with Objective 1 via test-retest, the investigators will then determine the limits of agreement between testing using SPNVT and ICNVT for patients known to have eye abnormalities that meet the inclusion/exclusion criteria. The first hypothesis is that testing using the SPNVT will be within a 95% limit of agreement with testing using ICNVT. The second hypothesis is that SPNVT will be non-inferior to ICNVT.
Primary Outcome Measure for Groups 7a and 7b | Study was conducted for each patient in one day.
  The The Test-Retest Repeatability for the identified three common near-vision procedures will be measured to determine sample sizes to reach the objectives of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa A Tang, MD, Principal Investigator — Neuro-ophthalmology of Texas
Locations (1):
- Neuro-ophthalmology of Texas, PLLC, Bellaire, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
After FDA decision will send our results and statistical analysis to an appropriate journal for publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: If FDA approval we will publish this data
Access Criteria: Access all of the above after publication